CLINICAL TRIAL: NCT00139009
Title: Intracellular and Renal/Myocardial Tissue Concentrations of Cyclosporine A (CsA) and Rejection Frequency Following Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oslo School of Pharmacy (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SUPER-CsA
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2007-06-15 (Estimated); Status verified 2006-09

CONDITIONS: Renal Transplantation; Heart Transplantation
Keywords: intracellular concentration; cyclosporine A; renal biopsies; heart biopsies; Renal transplant recipients
MeSH Terms: interventions — Cyclosporine

INTERVENTIONS:
Drug: Cyclosporine A

SUMMARY:
The primary objective is to investigate intralymphocyte concentrations of CsA in renal and heart transplant recipients to elucidate the association between the intracellular concentration and efficacy (rejection episodes and histology) in transplanted patients on CsA based immunosuppressive therapy.

DETAILED DESCRIPTION:
The primary objective is to investigate intralymphocyte concentrations of CsA in renal and heart transplant recipients to elucidate the association between the intracellular concentration and efficacy (rejection episodes and histology) in transplanted patients on CsA based immunosuppressive therapy.

Secondary objectives are to investigate associations between intralymphocyte concentrations and whole-blood concentrations of CsA, renal tissue concentrations and nephrotoxicity, heart tissue concentrations and cardiotoxicity with CsA based immunosuppressive therapy in transplanted patients. In addition, this study aims to validate the use of quinine as a probe for determination of CYP3A4 activity in transplanted patients as well as proteomic-based urine analyses as a screening tool for acute rejection episodes in transplanted patients.

ELIGIBILITY:
Inclusion Criteria:

1. Renal or heart transplant recipients scheduled to receive CsA as part of their immunosuppressive therapy at the time of transplantation.
2. 18 years of age or older.
3. Signed informed consent.

Exclusion Criteria:

1. Known contraindications for renal or heart biopsies, respectively, at the time of inclusion.
2. Concomitant treatment with: diltiazem, verapamil, phenytoin, carbamazepine, fluconazole, ketoconazole, erythromycin, clarithromycin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-06; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
rejection
pharmacokinetics

SECONDARY OUTCOMES:
toxicity
genotypes
metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Anders Åsberg, MSc, Study Director — University of Oslo
Locations (1):
- Rikshospitalet, Section of Nephrology, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Loftheim H, Midtvedt K, Hartmann A, Reisaeter AV, Falck P, Holdaas H, Jenssen T, Reubsaet L, Asberg A. Urinary proteomic shotgun approach for identification of potential acute rejection biomarkers in renal transplant recipients. Transplant Res. 2012 Aug 31;1(1):9. doi: 10.1186/2047-1440-1-9. PMID 23369437